CLINICAL TRIAL: NCT07292402
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics/Pharmacodynamics, and Antitumor Activity of JSKN022 in Subjects With Advanced Malignant Solid Tumors
Brief Title: JSKN022 in Subjects With Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JSKN022-101
Record Dates: First submitted 2025-11-13; First posted 2025-12-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: JSKN022; PD-L1; ITGB6; Antibody-Drug Conjugates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Dose escalation cohorts 1 (Experimental)
  Interventions: Drug: JSKN022
- Dose escalation cohort 2 (Experimental)
  Interventions: Drug: JSKN022
- Dose escalation cohort 3 (Experimental)
  Interventions: Drug: JSKN022
- Dose escalation cohort 4 (Experimental)
  Interventions: Drug: JSKN022
- Dose escalation cohort 5 (Experimental)
  Interventions: Drug: JSKN022
- Dose escalation cohort 6 (Experimental)
  Interventions: Drug: JSKN022
- Dose escalation cohort 7 (Experimental)
  Interventions: Drug: JSKN022
- Dose escalation cohort 8 (Experimental)
  Interventions: Drug: JSKN022
- Dose optimization cohort in selected tumor type 1 (Experimental)
  Interventions: Drug: JSKN022
- Dose optimization cohort in selected tumor type 2 (Experimental)
  Interventions: Drug: JSKN022
- Dose optimization cohort 3 - other advanced epithelial malignant tumors cohort (Experimental)
  Interventions: Drug: JSKN022

INTERVENTIONS:
Drug: JSKN022 — JSKN022 administered intravenously at selected dose levels according to protocol

SUMMARY:
The goal of this clinical trial is to learn if drug JSKN022 is safe to treat patients with advanced malignant solid tumors. It will also learn about the pharmacokinetic/ pharmacodynamic profiles and preliminary antitumor activity of drug JSKN022.

DETAILED DESCRIPTION:
This is a Phase I, open-label, multi-center, first-in-human (FIH) clinical trial designed to evaluate the safety, tolerability, pharmacokinetic (PK)/pharmacodynamic (PD) profiles, and antitumor activity of JSKN022 in patients with advanced malignant solid tumors.

Patients to be enrolled are with advanced unresectable or metastatic epithelial-derived malignant solid tumors confirmed by histology and/or cytology, who have failed previous standard treatment (disease progression), or be intolerant to standard treatment, or have no access to standard treatment.

The primary objective of the study is to evaluate the safety and tolerability of JSKN022 in patients with advanced malignant solid tumors and to determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) of JSKN022.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign the informed consent form.
2. Age ≥ 18 years old, male or female.
3. Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
4. Expected survival ≥ 3 months.
5. Histologically or cytologically confirmed malignant solid tumors confirmed by histology and/or cytology, who have failed previous standard treatment (disease progression), are intolerant to standard treatment, or have no access to standard treatment.
6. At least one measurable lesion at baseline according to RECIST 1.1 criteria.
7. Adequate organ function.
8. Agree to provide Recently archived or fresh tumor tissue samples.
9. Female subjects of childbearing potential or male subjects whose partners are of childbearing potential agree to use effective contraceptive measures.
10. Female subjects of childbearing potential must have a negative serum/urine pregnancy test within 7 days before the first dose.
11. Be able and willing to comply with the visits, treatment plans, laboratory tests, and other study-related procedures specified in the study protocol.
12. Adequate washout period of previous therapy before the first dose.

Exclusion Criteria:

1. Complicated with other malignant tumors within 5 years before the first dose, except for tumor types that have achieved clinical cure through local treatment with extremely low recurrence risk or tumor types with disease-free survival ≥ 5 years after radical treatment and extremely low recurrence/metastasis risk.
2. History of brainstem, meningeal metastasis, spinal cord metastasis or compression, or carcinomatous meningitis; presence of active brain metastasis.
3. Screening imaging shows tumor invasion, compression, or occurrence in surrounding important organs or risk of esophagotracheal fistula or esophagopleural fistula, except those judged by the investigator and medical monitor to not affect the patient's enrollment and administration.
4. Presence of clinically severe respiratory impairment caused by pulmonary disease complications.
5. Presence of the risk factors related to interstitial lung disease (ILD) or non-infectious pneumonia:
6. Presence of cardiovascular and cerebrovascular diseases or cardiovascular and cerebrovascular risk factors.
7. Gastrointestinal abnormalities with obvious clinical manifestations.
8. Active autoimmune diseases requiring systemic treatment within the past two years.
9. Significant serous effusion.
10. Uncontrolled infection.
11. Require regular glucocorticoid or immunosuppressive therapy.
12. Received live vaccines within 28 days before the first dose, or plan to receive live vaccines during the study period.
13. Prior treatment with antibody-drug conjugates containing topoisomerase I inhibitors.
14. Previous occurrence of grade ≥ 3 immune-related adverse events during immunotherapy.
15. Toxicity of previous anti-tumor treatment has not fully or partially recovered.
16. Known allergy to any component of the study drug, or history of severe allergic reactions to other antibody drugs.
17. Pregnant and/or lactating women, or planning to become pregnant during the study period.
18. Known history of mental illness, substance abuse, alcoholism, etc., or other situations that the investigator deems may affect the safety or compliance of the study drug treatment.
19. Local or systemic diseases caused by non-malignant tumors, or diseases or symptoms secondary to tumors, which may lead to high medical risks and/or uncertainty in survival assessment, such as tumor-related leukemia reaction (white blood cell count > 20×10⁹/L), cachexia manifestations, etc.
20. Any other previous or current diseases, treatments, or laboratory test abnormalities that the investigator deems may confuse the study results, affect the patient's full participation in the study, or participation in the study may not be in the best interest of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), serious adverse events (SAEs), etc (Safety and tolerability of JSKN-022). | From the first dose to 30 days after the last dose or until initiation of new anti-tumor treatment, whichever comes first.
  Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), serious adverse events (SAEs), etc.; abnormalities in physical examinations, laboratory tests, electrocardiograms, and other safety assessments.
Incidence of dose-limiting toxicity (DLT) in each dose group | 21 days from the first dose
Maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of JSKN022. | Up to 24 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | From the first study drug dose, until: disease progression per RECIST 1.1; initiation of new anti-tumor treatment; withdrawal of informed consent; death; loss to follow-up; or study termination, whichever comes first. Assessed at approximately 12 months.
  The proportion of subjects who achieve confirmed complete response (CR) or partial response (PR) as assessed by RECIST v1.1. ORR analysis will be based on the EAS set, with the proportion of subjects achieving objective response and the Clopper-Pearson exact 95% CI calculated.
Duration of response (DoR) | From the first study drug dose, until: disease progression per RECIST 1.1; initiation of new anti-tumor treatment; withdrawal of informed consent; death; loss to follow-up; or study termination, whichever comes first. Assessed up to 24 months.
  Defined as the time from the first documented evidence of response (PR or CR) to the first documented evidence of progressive disease (PD) or death from any cause in subjects with confirmed response (RECIST v1.1, PR or CR). For subjects without documented progression or death, DoR will be censored at the time of the last adequate tumor assessment. DoR analysis will be performed on subjects achieving CR or PR, with the median duration of response and 95% CI estimated using the Kaplan-Meier method.
Disease control rate (DCR) | From the first study drug dose, until: disease progression per RECIST 1.1; initiation of new anti-tumor treatment; withdrawal of informed consent; death; loss to follow-up; or study termination, whichever comes first. Assessed at approximately 12 months.
  The proportion of subjects who achieve confirmed CR, PR, or SD as assessed by RECIST v1.1. DCR analysis will be based on the EAS set, with the proportion of subjects achieving disease control and the Clopper-Pearson exact 95% CI calculated.
Clinical benefit rate (CBR) | From the first study drug dose, until: disease progression per RECIST 1.1; initiation of new anti-tumor treatment; withdrawal of informed consent; death; loss to follow-up; or study termination, whichever comes first. Assessed at approximately 12 months.
  The proportion of subjects who achieve confirmed CR, PR, or stable disease (SD) lasting more than 6 months as assessed by RECIST v1.1. CBR analysis will be based on the EAS set, with the proportion of subjects achieving clinical benefit and the Clopper-Pearson exact 95% CI calculated.
Progression-Free Survival (PFS) | From the first study drug dose, until: disease progression per RECIST 1.1; initiation of new anti-tumor treatment; withdrawal of informed consent; death; loss to follow-up; or study termination, whichever comes first. Assessed up to 24 months.
  Defined as the time from the first administration of the study drug to the first documentation of PD or death from any cause. PFS analysis will be based on the SAS set, with the median progression-free survival and 95% CI estimated using the Kaplan-Meier method. The 3-month, 6-month, 9-month, and 12-month progression-free survival rates and their 95% CIs will be calculated, and progression-free survival curves will be plotted.
6-Month and 12-Month Overall Survival Rates | From the first administration of the study drug until the death. Assessed up to 24 months.
  Defined as the probability of survival 6 months and 12 months after the first administration of the study drug, respectively. Analysis of 12-month survival rate will be based on the SAS set, with the 12-month survival rate and 95% CI estimated using the Kaplan-Meier method.
Incidence of anti-drug antibodies (ADA), antibody titers, and incidence of neutralizing antibodies (Nab, if applicable). | Up to 24 months
Maximum concentration (Cmax) of JSKN022 | From the enrollment until the end of study. Assessed up to 24 months.
  Maximum concentration (Cmax) of JSKN022
Time to maximum concentration (Tmax) of JSKN022 | From the enrollment until the end of study. Assessed up to 24 months.
  Time to maximum concentration (Tmax) of JSKN022
Trough concentration (Ctrough) of JSKN022 | From the enrollment until the end of study. Assessed up to 24 months.
  Trough concentration (Ctrough) of JSKN022
Area under the concentration-time curve of JSKN022 | From the enrollment until the end of study. Assessed up to 24 months.
  Area under the concentration-time curve of JSKN022
Volume of distribution (V) of JSKN022 | From the enrollment until the end of study. Assessed up to 24 months.
  Volume of distribution (V) of JSKN022
Elimination half-life (t1/2) of JSKN022 | From the enrollment until the end of study. Assessed up to 24 months.
  Elimination half-life (t1/2) of JSKN022
Clearance (CL) of JSKN022 | From the enrollment until the end of study. Assessed up to 24 months.
  Clearance (CL) of JSKN022

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No